CLINICAL TRIAL: NCT00165984
Title: Influence of Genetic Polymorphisms on Ventricular Structure and Function in Patients With Single Ventricle Anatomy
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Paul M. Kirshbom, MD, Associate professor of surgery, Emory University
Other Study IDs: 599-2004
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Congenital Heart Disease
Keywords: cardiac; hypoplastic; pediatric; hypoplastic heart ventricle
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum.
Oversight: Data Monitoring Committee: No

SUMMARY:
There are many kids born with congenital heart disease. Some of these defects may lead to the formation of a single ventricle (the heart having only one pumping chamber). These children normally undergo a series of corrective surgeries to help overcome the problems of having just one ventricle. However there are some differences in how well the patients respond to the surgeries. In the adult population, studies have shown that there may be a genetic link that may be responsible for the differences in how patients respond. The investigators would like to study the pediatric population by looking for certain genetic markers in the patients' blood. They will also collect basic health information on each patient.

DETAILED DESCRIPTION:
In the United States, approximately 30,000 children are born with congenital heart disease every year. Between 1000 and 2000 of these children have some form of functional single ventricle anatomy, with variants of hypoplastic left heart syndrome (HLHS) comprising about half. Patients with functional single ventricle anatomy are born with a malformation that renders one of their ventricles unusable and surgically unrecoverable. In HLHS, for example, either the mitral or aortic valve can be absent or significantly stenotic, which is generally associated with marked hypoplasia of the left ventricle and the ascending aorta. Other common variants of single ventricle anatomy are tricuspid or pulmonary atresia, often associated with some degree of right ventricular hypoplasia, unbalanced atrioventricular defects, in which either ventricle can be unusable due to malposition of the interventricular septum, and the heterotaxy syndromes. All of these congenital cardiac anomalies, as well as several other less common variants, can be treated with a multi-stage surgical palliation that usually requires three surgical procedures during the first three years of life. At the completion of this series of palliative procedures the children are left with their single functional ventricle driving blood flow to the systemic circulation while their pulmonary circulation is derived from passive drainage of the systemic venous return into and through the pulmonary vasculature. This arrangement, the so-called "Fontan physiology", can provide an excellent quality of life as these children grow and enter young adulthood; however, it is by no means a normal hemodynamic arrangement and a significant percentage of children with single ventricle anatomy will fail either during the early palliative steps or at some point after they achieve final Fontan palliation.

Failure of single ventricle patients to progress through the multi-stage palliation or late failure of patients after the Fontan procedure can result from a myriad of causes. While ventricular dysfunction is a common finding in failing single ventricle patients, an anatomic reason for their clinical failure, such as myocardial ischemia or ventricular outflow obstruction, often cannot be identified. Many of these patients subsequently die or require cardiac transplantation when their single ventricle fails. Because patient outcomes are highly variable despite similar anatomy and hemodynamics, it has been suggested that genetic variability may play a role in the ability of patients to tolerate long-term single ventricle palliation.

The interaction between genetic variability and outcomes has been well documented for adult patients with cardiovascular disease. Genetic polymorphisms in the renin-angiotensin system (RAS) in particular have been well studied. The active final product of the RAS is angiotensin-II, which is produced by the sequential cleavage of angiotensinogen (AGT) by renin and angiotensin-converting enzyme (ACE). Several steps in this series of enzymatic reactions have been evaluated as candidate genes of influence for cardiovascular disorders.

Polymorphisms in the AGT gene have been associated with essential hypertension, however, a subsequent study failed to demonstrate any influence of these polymorphisms on outcome in patients with idiopathic dilated cardiomyopathy. A polymorphism in the ACE gene involving a 287-base pair insertion (I) or deletion (D) has been evaluated in several studies. The DD genotype is associated with higher serum levels of ACE and angiotensin II, increased incidence of sudden death in patients with hypertrophic cardiomyopathy, increased mortality in patients with idiopathic heart failure, and decreased exercise tolerance in patients with congestive heart failure. Meanwhile, a genetic variant in the Angiotensin II type 2-receptor (AT2-R) has been shown to influence left ventricular structure and function in young men with hypertension.

Another potentially important contributor to ventricular function that has been studied with regard to genetic polymorphism related variability is the Beta1-adrenergic receptor (Beta1-AR). The Beta1-AR is the primary myocardial receptor for the catecholamines epinephrine and norepinephrine, which increase myocardial contractility and blood pressure. Several polymorphisms in the Beta1-AR gene have been associated with an increased risk for congestive heart failure and with exercise capacity in patients with ischemic or idiopathic cardiomyopathy.

A final area of interest is the opposing system of vasodilators and vasoconstrictors that control systemic vascular tone. Two major contributors to vasomotor tone in humans are the endothelium derived vasodilator nitric oxide (NO) and the powerful vasoconstrictor endothelin-1. Endothelial NO is produced by the enzyme endothelial nitric oxide synthase (eNOS). A single base-pair polymorphism (G894T) is associated with an increased risk of vasospastic angina pectoris and with increased vascular responsiveness to phenylephrine in patients on cardiopulmonary bypass. Meanwhile, a single base-pair polymorphism in the preproendothelin-1 (pp-ET1) gene (G5665T) has been shown to increase vasomotor reactivity in human mammary arteries. This polymorphism is also associated with hypertension in overweight patients with the T allele.

While there is very little data available regarding the causes of failure in children with single ventricle anatomy, it is clear that genetic factors which influence ventricular function and the development of heart failure in adults with two ventricles could play a role in the failure of patients with one ventricle. We propose a combined retrospective and prospective evaluation of each of the candidate gene polymorphisms discussed above for potential linkage to poor outcome in children with single ventricle anatomy. Poor outcome for these children would be defined as a multi-endpoint variable including death, evaluation for heart transplantation, or the development of severe single ventricle dysfunction by echocardiographic or cardiac catheterization criteria. Identification of high-risk combinations of genetic alleles could guide therapy for patients with poor predicted outcome, possibly steering such patients towards early transplantation rather than attempted staged palliation.

ELIGIBILITY:
Inclusion Criteria:

* Children who currently have functional single ventricle anatomy or have had heart transplantation for single ventricle anatomy who receive their cardiac care at Children's Healthcare of Atlanta, Egleston Hospital.
* Family agrees to participate in the study following informed consent

Exclusion Criteria:

* Conversion to two ventricle physiology, excluding transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pediatric single ventricle patients or pediatric patients previously transplanted for single ventricle, who undergo an invasive procedure (surgery or catheterization) will be a candidate for enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2004-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Kirshbom, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Marian AJ, Yu QT, Workman R, Greve G, Roberts R. Angiotensin-converting enzyme polymorphism in hypertrophic cardiomyopathy and sudden cardiac death. Lancet. 1993 Oct 30;342(8879):1085-6. doi: 10.1016/0140-6736(93)92064-z. PMID 8105312
- [Background] Small KM, Wagoner LE, Levin AM, Kardia SL, Liggett SB. Synergistic polymorphisms of beta1- and alpha2C-adrenergic receptors and the risk of congestive heart failure. N Engl J Med. 2002 Oct 10;347(15):1135-42. doi: 10.1056/NEJMoa020803. PMID 12374873
- [Background] Iglarz M, Benessiano J, Philip I, Vuillaumier-Barrot S, Lasocki S, Hvass U, Durand G, Desmonts JM, Levy BI, Henrion D. Preproendothelin-1 gene polymorphism is related to a change in vascular reactivity in the human mammary artery in vitro. Hypertension. 2002 Feb;39(2):209-13. doi: 10.1161/hy0202.103442. PMID 11847185
- [Background] Wagoner LE, Craft LL, Zengel P, McGuire N, Rathz DA, Dorn GW 2nd, Liggett SB. Polymorphisms of the beta1-adrenergic receptor predict exercise capacity in heart failure. Am Heart J. 2002 Nov;144(5):840-6. doi: 10.1067/mhj.2002.125325. PMID 12422153

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Ventricle Patients: Patients born with single ventricle heart disease
Period: Overall Study
Arm/Group | Single Ventricle Patients
Started | 165
Completed | 150
Not Completed | 15
Not completed — Death | 15

BASELINE CHARACTERISTICS:
Arm/Group | Single Ventricle Patients
Number analyzed (Participants) | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 165
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 108
Region of Enrollment [Number; unit: participants]
  United States | 165

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Incidence of the Pre-proendothelin SNP at Nucleotide 5665
Time Frame: 7 years
Population: 165 enrolled patients were analyzed for this polymorphism
Measure: Number; unit: participants
Groups:
- Incidence of Preproendothelin-1 5665 Polymorphism: Incidence of Homozygosity for mutation at nucleotide 5665
Arm/Group | Incidence of Preproendothelin-1 5665 Polymorphism
Number analyzed (Participants) | 165
participants | 10

2. Primary Outcome: Survival
Description: Follow-up study designed to determine the impact of genetic factors on survival in single ventricle patients
Time Frame: 7 yr mean follow-up
Population: All patients enrolled were genotyped
Measure: Number; unit: percentage of patients alive/nontrans
Groups:
- Preproendothelin-1 (ppET1) 5665 Polymorphism Homozygotes: Transplant-free survival for patients homozygous for T at nucleotide 5665 at 7 years.
- Homozygous for Wild-type ppET1 5665: Transplant-free survival for patients homozygous for G at nucleotide 5665 at 7 years.
- Heterozygotes: Transplant-free survival for patients heterozygous (G/T) at nucleotide 5665 at 7 years.
Arm/Group | Preproendothelin-1 (ppET1) 5665 Polymorphism Homozygotes | Homozygous for Wild-type ppET1 5665 | Heterozygotes
Number analyzed (Participants) | 10 | 103 | 52
percentage of patients alive/nontrans | 40 [10 to 10] | 80 | 88
Statistical Analysis 1: Comparison: Preproendothelin-1 (ppET1) 5665 Polymorphism Homozygotes vs Homozygous for Wild-type ppET1 5665 vs Heterozygotes; Test type: Superiority or Other; p = 0.003, Regression, Cox; Odds Ratio (OR) = 4.9, 95% CI 2-sided [1.7 to 13.9]

ADVERSE EVENTS:
Arm/Group | Single Ventricle Patients
Serious Adverse Events (participants affected / at risk) | 0/165
Other Adverse Events (participants affected / at risk) | 0/165

LIMITATIONS AND CAVEATS:
Relatively small number of patients given the low incidence of this mutation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No